CLINICAL TRIAL: NCT04502953
Title: Outcome of Vertical Versus Horizontal Plicataion in Transperienal Repair of Rectocele; a Randomized Controlled Trial
Brief Title: Vertical Versus Horizontal Plicataion in Transperienal Repair of Rectocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mansoura20201
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Rectocele
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vertical plication (Active Comparator): Vertical plication of the rectovaginal septum was done
  Interventions: Procedure: Vertical plication
- Horizontal plication (Active Comparator): Horizontal plication of the rectovaginal septum was done
  Interventions: Procedure: Horizontal plication

INTERVENTIONS:
Procedure: Vertical plication — Vertical plication of the rectovaginal septum was done
  Arms: Vertical plication
Procedure: Horizontal plication — Horizontal plication of the rectovaginal septum was done
  Arms: Horizontal plication

SUMMARY:
We assumed that the technique of plication of the rectovaginal septum and rectal wall may factor in providing better and more sustained repair that confers more satisfactory improvement in symptoms. The present randomized study aimed to evaluate the outcome of TPR with vertical plication of the rectovaginal septum as compared to the horizontal plication with regards to improvement in ODS, recurrence of rectocele, postoperative complications and dyspareunia.

ELIGIBILITY:
Inclusion Criteria:

* Vertical plication of the rectovaginal septum was done

Exclusion Criteria:

* patients with ODS caused by conditions other than rectocele such as anismus and internal rectal prolapse
* patients with slow transit constipation.
* patients with recurrent rectocele after previous surgery.
* patients with pre-existing FI
* patients with associated anorectal pathology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Complete cure of symptoms | 12 months after repair
  Absence of symptoms of constipation with Wexner score <2

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, Study Chair — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided